CLINICAL TRIAL: NCT03302091
Title: Pharmacokinetics, Safety and Tolerability After Multiple Dose Administration of BI 1467335 in Subjects With Moderate Renal Impairment and Subjects With Normal Renal Function (a Mono-centric, Open-label Study in Matched-group Design)
Brief Title: A Study in People With Normal Kidney Function and People With Reduced Kidney Function to Test How BI 1467335 is Processed in the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1386-0002; 2017-002180-18 (EudraCT Number)
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Results first posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Renal Insufficiency; Healthy
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 1467335 Normal (R) (Experimental): Participants with normal renal function.
  Interventions: Drug: BI 1467335
- BI 1467335 Moderate (T) (Experimental): Participants with moderate renal impairment.
  Interventions: Drug: BI 1467335

INTERVENTIONS:
Drug: BI 1467335 — 28 day treatment period

SUMMARY:
The primary objective of the current study is to investigate the influence of moderate renal impairment on the pharmacokinetics of multiple doses in comparison to a matched control group with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Despite of moderate renal impairment (Group 1) healthy male or female subjects according to the assessment of the investigator, based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Estimated glomerular filtration rate (eGFR) based on CKD-EPI formula for Group 1 between 30 and 59 mL/min/1.73m2 and for Group 2 ≥ 90 mL/min/1.73m2
* Age of 18 to 79 years (incl.)
* BMI of 18.5 to 34 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation
* Male subjects, or female subjects who meet any of the following criteria (according to the CTFG Recommendations related to contraception and pregnancy testing in clinical trials, methods with a failure rate of less than 1% per year) starting from at least 30 days before the first administration of trial medication and until 30 days after trial completion, e.g.:

  * Use of adequate contraception, e.g. any of the following methods plus condom: implants, injectables, combined oral or vaginal contraceptives (inhibition of ovulation)
  * Hormonal intrauterine device
  * Sexually abstinent (defined as refraining from heterosexual intercourse during the entire period of risk)
  * A vasectomised sexual partner (provided that vasectomy was performed at least 1 year prior to enrolment and the vasectomised partner has received medical assessment of the surgical success)
  * Surgically sterilised (including bilateral tubal occlusion, hysterectomy)
  * Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous levels of FSH above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

Healthy subjects

* Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Estimated glomerular filtration rate (eGFR) calculated by CKD-EPI formula < 90 mL/min/1.73m2

Subjects with moderate renal impairment

* Subject with significant diseases other than moderate renal impairment. A significant disease is defined as a disease which in the opinion of the investigator:

  * puts the subjects at risk because of participation in the study
  * may influence the results of the study
  * may influence the subject's ability to participate in the study
  * is not in a stable condition Diabetic or hypertensive subjects can be entered in this trial if the disease is not significant according to these criteria.
* Any finding of the medical examination (including BP, PR and ECG) of clinical relevance
* Moderate and severe concurrent liver function impairment (e.g. due to hepatorenal syndrome) or biliary obstruction
* Clinically relevant laboratory abnormalities (except for renal function tests or deviation of clinical laboratory values that are related to renal impairment)
* eGFR calculated by CKD-EPI formula ≥ 60 mL/min/1.73m2 and < 30 mL/min/1.73m2

For all subjects

* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 30 days prior to planned administration of trial medication or longer if required by local regulation, or within 5-half-lives of the investigational agent taken (whichever is longer), or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 20 g per day for females and 30 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males or repeatedly greater than 470 ms in females) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

Female subjects will not be allowed to participate if any of the following applies:

* Positive pregnancy test, pregnancy or plans to become pregnant within 30 days after study completion
* Lactation period

Male subjects will not be allowed to participate if any of the following applies:

- Male subjects with WOCBP partner who are unwilling to use male contraception (condom or sexual abstinence) from the first administration of trial medication until 30 days after last administration of trial medication

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2018-08-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Kiel GmbH, Kiel, Germany

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was open-label, multiple-dose and matched-group design. 20 participants entered (ten in each of the two groups). Participants with moderate renal impairment were assigned to the moderate group and individually matched participants with normal renal function were assigned to the normal group.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended a specialist site which would then ensure that they (the participants) met all strictly implemented inclusion/exclusion criteria. Participants were not to be assigned to treatment groups if any one of the specific entry criteria were violated.
Groups:
- BI 1467335 Normal (R): Participants with normal renal function were administered 10 milligram (mg) (5 mg X2) BI 1467335 film coated tablet orally with 240 milliliter (mL) water after an overnight fast of at least 10 hour (h) once daily over 28 days.
- BI 1467335 Moderate (T): Participants with moderate renal impairment were administered 10 milligram (mg) (5 mg X2) BI 1467335 film coated tablet orally with 240 milliliter (mL) water after an overnight fast of at least 10 hour (h) once daily over 28 days.
Period: Overall Study
Arm/Group | BI 1467335 Normal (R) | BI 1467335 Moderate (T)
Started (Started are treated) | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The TS included all subjects who were documented to have taken at least one dose of trial medication. This is the full analysis set population in the sense of International council for harmonisation - efficacy guideline 9: statistical principles for clinical trials (ICH-E9).
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 1467335 Normal (R) | BI 1467335 Moderate (T) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.5 (9.5) | 68.7 (10.9) | 68.1 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 1467335 in Plasma Over the Time Interval From 0 to 24 Hours After Administration of the First Dose (AUC0-24)
Description: Area under the concentration-time curve of BI 1467335 in plasma over the time interval from 0 to 24 hours after administration of the first dose AUC 0-24.
  Standard Error presented is actually geometric Standard Error. PKS-stat including participants data for AUC(0-24). The pharmacokinetic (PK) analysis set (PKS) included all subjects in the TS who provided at least one PK parameter that was defined as primary or secondary endpoint and who were not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Time Frame: Pharmacokinetic (PK) samples were taken 2.00 hours (h) before dosing and 0.25, 0.50, 0.75, 1.00, 1.50, 2.00, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00 and 23.917 h after dosing on day 1.
Population: PK statistical analysis set (PKS-stat) included all subjects from PK set who built a subject pair of renally impaired subject and her/his matching healthy volunteer control and provided at least one primary or secondary PK parameter and who were not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole*hour/Liter (nmol*h/L)
Arm/Group | BI 1467335 Normal (R) | BI 1467335 Moderate (T)
Number analyzed (Participants) | 9 | 9
nanomole*hour/Liter (nmol*h/L) | 3.97 (1.31) | 7.88 (1.31)
Statistical Analysis 1: Comparison: BI 1467335 Normal (R) vs BI 1467335 Moderate (T); The statistical model used for the analyses of the primary endpoints was an ANOVA (analysis of variance) model on the logarithmic scale including the effect "degree of renal impairment" as a fixed effect as well as subject pair as a random effect; Test type: Other; ANOVA; Adjusted gMean ratio (T/R)% = 198.50, 90% CI 2-sided [101.83 to 386.94], Standard Deviation 96.5 — Standard deviation is actually intra individual geometric coefficient of variation (%)

2. Primary Outcome: Maximum Measured Concentration of BI 1467335 in Plasma After Administration of the First Dose (Cmax)
Description: Maximum measured concentration of BI 1467335 in plasma after administration of the first dose (Cmax).
  Standard Error presented is actually geometric Standard Error.
Time Frame: Pharmacokinetic (PK) samples were taken 2.00 h before dosing and 0.25, 0.50, 0.75, 1.00, 1.50, 2.00, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00 and 23.917 h after dosing on day 1.
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole/Liter (nmol/L)
Arm/Group | BI 1467335 Normal (R) | BI 1467335 Moderate (T)
Number analyzed (Participants) | 10 | 10
nanomole/Liter (nmol/L) | 3.03 (1.24) | 6.01 (1.24)
Statistical Analysis 1: Comparison: BI 1467335 Normal (R) vs BI 1467335 Moderate (T); [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Adjusted gMean ratio (T/R)% = 198.42, 90% CI 2-sided [116.56 to 337.78], Standard Deviation 77.5 — Standard deviation is actually intra individual geometric coefficient of variation (%)

3. Primary Outcome: Area Under the Concentration-time Curve of BI 1467335 in Plasma Over the Dosing Interval After Administration of the 28th Dose (AUCτ,28)
Description: Area under the concentration-time curve of BI 1467335 in plasma over the dosing interval after administration of the 28th dose (AUCτ,28).
  Standard Error presented is actually geometric Standard Error. As per the protocol, day is counted as "Day 1 = 0:00".
Time Frame: Pharmacokinetic samples were taken 0.0833 h before last dose and 0.25, 0.50, 0.75, 1.00, 1.50, 2.00, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00 and 24.00 h after dosing on day 28.
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole*hours/Liter (nmol*h/L)
Arm/Group | BI 1467335 Normal (R) | BI 1467335 Moderate (T)
Number analyzed (Participants) | 10 | 10
nanomole*hours/Liter (nmol*h/L) | 692.42 (1.23) | 1566.88 (1.23)
Statistical Analysis 1: Comparison: BI 1467335 Normal (R) vs BI 1467335 Moderate (T); [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Adjusted gMean ratio (T/R)% = 226.29, 90% CI 2-sided [156.35 to 327.53], Standard Deviation 47.5 — Standard deviation is actually intra individual geometric coefficient of variation (%)

4. Primary Outcome: Maximum Measured Concentration of BI 1467335 in Plasma Following Administration of the 28th Dose (Cmax,28)
Description: Maximum measured concentration of BI 1467335 in plasma following administration of the 28th dose (Cmax,28).
  Standard Error presented is actually geometric Standard Error. As per the protocol, day is counted as "Day 1 = 0:00".
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole/Liter (nmol/L)
Arm/Group | BI 1467335 Normal (R) | BI 1467335 Moderate (T)
Number analyzed (Participants) | 10 | 10
nanomole/Liter (nmol/L) | 100.57 (1.13) | 141.20 (1.13)
Statistical Analysis 1: Comparison: BI 1467335 Normal (R) vs BI 1467335 Moderate (T); [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Adjusted gMean ratio (T/R)% = 140.40, 90% CI 2-sided [108.06 to 182.43], Standard Deviation 32.8 — Standard deviation is actually intra individual geometric coefficient of variation (%)

5. Secondary Outcome: Area Under the Concentration-time Curve of BI 1467335 in Plasma Over the Dosing Interval After Administration of the 14th Dose (AUCτ,14)
Description: Area under the concentration-time curve of BI 1467335 in plasma over the dosing interval after administration of the 14th dose (AUCτ,14).
  Standard Error presented is actually geometric Standard Error. As per the protocol, day is counted as "Day 1 = 0:00".
Time Frame: Pharmacokinetic samples were taken 0.0833 h before dosing and 0.25, 0.50, 0.75, 1.00, 1.50, 2.00, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00 and 23.917 h after dosing on day 14.
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole*hour/Liter (nmol*h/L)
Arm/Group | BI 1467335 Normal (R) | BI 1467335 Moderate (T)
Number analyzed (Participants) | 10 | 10
nanomole*hour/Liter (nmol*h/L) | 321.23 (1.34) | 532.06 (1.34)
Statistical Analysis 1: Comparison: BI 1467335 Normal (R) vs BI 1467335 Moderate (T); [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Adjusted gMean ratio (T/R)% = 165.63, 90% CI 2-sided [107.51 to 255.17], Standard Deviation 56.6 — Standard deviation is actually intra individual geometric coefficient of variation (%)

6. Secondary Outcome: Maximum Measured Concentration of BI 1467335 in Plasma Following Administration of the 14th Dose (Cmax,14)
Description: Maximum measured concentration of BI 1467335 in plasma following administration of the 14th dose (Cmax,14).
  Standard Error presented is actually geometric Standard Error. As per the protocol, day is counted as "Day 1 = 0:00".
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole/Liter (nmol/L)
Arm/Group | BI 1467335 Normal (R) | BI 1467335 Moderate (T)
Number analyzed (Participants) | 10 | 10
nanomole/Liter (nmol/L) | 73.41 (1.16) | 94.28 (1.16)
Statistical Analysis 1: Comparison: BI 1467335 Normal (R) vs BI 1467335 Moderate (T); [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Adjusted gMean ratio (T/R)% = 128.44, 90% CI 2-sided [99.64 to 165.57], Standard Deviation 31.7 — Standard deviation is actually intra individual geometric coefficient of variation (%)

ADVERSE EVENTS:
Time Frame: From first day of study drug administration until End of trial (EOT), up to 41 days.
Description: The treated set (TS) included all subjects who were documented to have taken at least one dose of trial medication. This is the full analysis set population in the sense of ICH-E9.
Arm/Group | BI 1467335 Normal (R) | BI 1467335 Moderate (T)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/10 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1467335 Normal (R) (N=10) | BI 1467335 Moderate (T) (N=10)
Vomiting (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT03302091/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT03302091/SAP_001.pdf